CLINICAL TRIAL: NCT04914364
Title: Describing Balance Function in Patients Post-COVID-19
Brief Title: Balance Function in Patients Post Corona Virus Disease 2019 (COVID-19)
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00108353
Record Dates: First submitted 2021-06-02; First posted 2021-06-04 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Covid19
Keywords: COVID; Balance
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have tested positive for COVID-19: Patients who are designated as "COVID recovered" in the electronic medical record and who fit the inclusion criteria.
  Interventions: Other: Balance assessments

INTERVENTIONS:
Other: Balance assessments — There is no formal intervention in this study. The investigators will only be completing balance assessments with no follow-up visit.

SUMMARY:
The purpose of this study is to describe balance deficits in patients post COVID-19. The information the investigators learn may help influence balance training exercises for patients post-COVID-19. Participants will have a primary or secondary diagnosis of COVID-19 during hospitalization and off COVID-19 isolation and be receiving care in an acute inpatient hospital. Following consent, participants will complete balance assessments and questionnaires about balance and dizziness in a single session. Vital signs will be monitored during the session.The greatest risks of this study include shortness of breath, and a risk of falling or musculoskeletal soreness.These risks are no greater than those experienced during a usual physical therapy visit.

DETAILED DESCRIPTION:
Heart rate (HR), respiratory rate (RR), blood pressure (BP), and oxygen saturation (SpO2) will be measured at rest and after all outcome measures are completed. Rate of Perceived Exertion (RPE) (0-10 per modified Borg scale) will be measured after each outcome measure. In addition, HR will be measured after each outcome measure. SpO2 will be continually monitored via pulse oximetry. Fraction of inspired oxygen (FiO2) will be titrated per MD orders. If SpO2 drops below MD-specified parameters, patients will first be given a 3-minute seated rest break. If SpO2 recovers above MD-specified parameters after rest break, activity will resume. If SpO2 remains below MD-specified parameters after rest break or continues to drop with activity, FiO2 will be titrated to maintain SpO2 within MD-specified parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Primary or secondary diagnosis of COVID- 19 during hospitalization and off COVID-19 isolation
* Receiving care in acute inpatient
* Ability to ambulate 20' with or without an assistive device without dropping >10% of resting oxygen saturation (determined from existing physical therapy evaluation)
* Ability to stand with no more than contact guard assistance (determined from existing physical therapy evaluation)
* Not requiring use of mechanical ventilation
* Minimum resting oxygen saturation of 88% with or without supplemental oxygen
* No neurological or orthopedic dysfunction that would affect balance
* Cognitively intact and able to follow directions and provide consent

Exclusion Criteria:

* History of 2 or more falls in the year prior to COVID-19 diagnosis or history of balance dysfunction

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects will be adults who have primary or secondary diagnosis of COVID-19 during hospitalization and off COVID-19 isolation and be receiving care in an acute inpatient hospital (Duke University Health System).
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Poole, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from a large academic medical center.
Period: Overall Study
Arm/Group | Patients Who Have Tested Positive for COVID-19
Started | 28
Completed | 25
Not Completed | 3
Not completed — No longer eligible for study | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Arm/Group | Patients Who Have Tested Positive for COVID-19
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25
Resting FiO2 [Mean (Standard Deviation); unit: percentage of inspired oxygen] — The fraction of inspired oxygen (FiO2) is an estimation of the oxygen content a person inhales.
  percentage of inspired oxygen | 1.04 (2.07)
Resting SpO2 [Mean (Standard Deviation); unit: percentage of oxygen-saturated blood] — SpO2 is the percentage of blood that is saturated with oxygen.
  percentage of oxygen-saturated blood | 96.92 (2.14)
Time since COVID diagnosis [Mean (Standard Deviation); unit: days] | 34.44 (15.35)

OUTCOME MEASURES:

1. Primary Outcome: Motor Balance as Measured by Timed Up and Go (TUG)
Description: The TUG measures mobility, motor balance, walking ability, and falls risk based on how long it takes the patient to stand up, walk 10 feet, turn around, walk back, and sit down. < 10 seconds = normal, < 20 seconds = good mobility; can walk outside alone; does not require a walking aid, < 30 seconds = walking and balance problems; cannot walk outside alone; requires walking aid.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Patients Who Have Tested Positive for COVID-19
Number analyzed (Participants) | 25
seconds | 20.57 (10.34)

2. Secondary Outcome: Sensory Influence on Balance as Measured by Modified Clinical Test of Sensory Interaction in Balance (mCTSIB)
Description: The mCTSIB assesses how well a patient is using sensory inputs when one or more sensory systems are compromised based on how long it takes the patient to complete the task under four different conditions. 1) Eyes Open, Firm Surface; 2) Eyes Closed, Firm Surface; 3) Eyes Open, Foam Surface; 4) Eyes Closed, Foam Surface. The trial is over when (a) the participant opens his/her eyes in an eyes closed condition, (b) raises arms from sides, (c) loses balance and requires manual assistance to prevent a fall.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Patients Who Have Tested Positive for COVID-19
Number analyzed (Participants) | 25
seconds
  mCTSIB eyes open firm surface | 30.0 (0.00)
  mCTSIB eyes closed firm surface | 28.28 (6.24)
  mCTSIB eyes open foam surface | 27.50 (8.08)
  mCTSIB eyes closed foam surface | 19.41 (1.89)

3. Secondary Outcome: Balance Confidence as Measured by Activities Specific Balance Confidence (ABC) Scale
Description: Self-report questionnaire where patients rate their balance confidence for performing activities. Scores range 0-100 where 0 indicates no balance confidence and 100 indicates complete balance confidence.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Who Have Tested Positive for COVID-19
Number analyzed (Participants) | 25
score on a scale | 66.88 (17.61)

ADVERSE EVENTS:
Time Frame: During a single study visit, up to 3 hours
Description: All assessments were performed during one study visit.
Arm/Group | Patients Who Have Tested Positive for COVID-19
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT04914364/Prot_SAP_000.pdf